CLINICAL TRIAL: NCT01999231
Title: Phase I Clinical Human Tolerability Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Air Force Military Medical University, China (Other); Proswell Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LTao-EC; LTao (Registry Identifier: AnhuiZhifei)
Record Dates: First submitted 2013-11-04; First posted 2013-12-03 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Safety; Tolerability; ESAT6; CFP10; skin test; diagnostic test
MeSH Terms: interventions — ESAT-6-CFP10 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1μg/ml ESAT6-CFP10 (Experimental): The 1μg/ml ESAT6-CFP10 is given 0.1ml alone to volunteers in the RIGHT or LEFT forearm according to a randomisation scheme.
  Interventions: Biological: ESAT6-CFP10
- 5μg/ml ESAT6-CFP10 (Experimental): The 5μg/ml ESAT6-CFP10 is given 0.1ml alone to volunteers in the RIGHT or LEFT forearm according to a randomisation scheme.
  Interventions: Biological: ESAT6-CFP10
- 10μg/ml ESAT6-CFP10 (Experimental): The 10μg/ml ESAT6-CFP10 is given 0.1ml alone to volunteers in the RIGHT or LEFT forearm according to a randomisation scheme.
  Interventions: Biological: ESAT6-CFP10
- 20μg/ml ESAT6-CFP10 (Experimental): The 20μg/ml ESAT6-CFP10 is given 0.1ml alone to volunteers in the RIGHT or LEFT forearm according to a randomisation scheme.
  Interventions: Biological: ESAT6-CFP10

INTERVENTIONS:
Biological: ESAT6-CFP10 — 32 healthy subjects who meet the standard of protocol are allocated four different groups according to dosages of ESAT6-CFP10 :1μg/ml ESAT6-CFP10、5μg/ml ESAT6-CFP10、10μg/ml ESAT6-CFP10、20μg/ml ESAT6-CFP10.Each dose group have six healthy subjects(three male and three female) , at the same time set up two people for substitute (one male and one female) . ESAT6-CFP10 administered intradermally by the mantoux injection technique. Each receives only one dosage in right or left arm .
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10; EC

SUMMARY:
In the tests, small sample of clinical study about Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 ( Recombination EC Allergen） healthy adults was carried out.

24 healthy adults were included as study objects, they were randomly divided into four groups of different Recombinant Allergen EC dose (1, 5, 10μg/mL, maximum tolerated dose 20μg/mL, 6 person/dose) for single arm intradermal injection.

The main examination items :vital signs (breathing, heart rate, blood pressure, body temperature ) of each volunteer at 15min, 30min, 1h, 2h, 4h, 8h, 24h, 48h, 72h, 96h after injection, skin reactivity (redness and/or induration) diameter of injection sites,local reaction ( rash, pain, itching, and skin and mucous membranes ) ,a variety of adverse events,routine blood,routine urine, liver and kidney function, ECG and chest X-ray films before and 7 days after intradermal injection .

Preliminary evaluation of safety and tolerability of Recombinant Allergen EC applied in humans, which can provide a safe dosage range for phase II clinical study.

DETAILED DESCRIPTION:
This clinical study adopts an open, randomized study methods to carry out Recombinant EC Allergen on small sample of healthy adults.

24 healthy adults were included as study objects, they were randomly divided into four groups of different Recombinant EC Allergen dose (1, 5, 10μg/mL, maximum tolerated dose 20μg/mL, 6 person/dose) for single arm intradermal injection, and set up two people as replacement for each group (one male and one female).

Intradermal injection into one third site of healthy subjects' left or right forearm palmaris with 0.1ml Recombinant EC Allergen for only one time.

The main examination items :vital signs (breathing, heart rate, blood pressure, body temperature ) of each volunteer at 15min, 30min, 1h, 2h, 4h, 8h, 24h, 48h, 72h, 96h after injection, skin reactivity (redness and/or induration) diameter of injection sites,local reaction ( rash, pain, itching, and skin and mucous membranes ) ,a variety of adverse events,routine blood,routine urine, liver and kidney function, ECG and chest X-ray films before and 7 days after intradermal injection .

In phaseⅠclinical study, each person can accept only one dose, After injection of the same dose of a volunteer group, be sure the next injection of a volunteer at 40 minutes interval. Different dose groups: the next dose test should be carried on in the case of no serious adverse events appear in 7days after the last one volunteer's injection in a former lower dose group.

Statistical analysis is performed using SAS9.3 software, and all analytic process is routinization.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 40 years old, age difference is not more than 10 years old within the same batch of healthy volunteers, the male to female ratio of cases is 1:1. Body mass index should be in the range of 20 to 27 Body Mass Index BMI: weight (Kg)/ height (M2);
* Agreed to participate in the test and sign the informed consent;
* Subjects should comply with the requirements of the clinical trial protocol and be followed;
* Subjects have no history of TB (Tuberculosis)or family history of tuberculosis;
* People have no pulmonary tuberculosis or extrapulmonary tuberculosis,respiratory symptom or systemic symptoms;
* People have no tuberculosis focus after examination by X-ray chest radiograph and sputum bacilli;
* Subjects have no acute or chronic disease, acute infectious diseases, dermatoses or skin allergy caused by various reasons;
* Physical condition: have no history of heart, liver, kidney, gastrointestinal tract, nervous system, or metabolic disturbance, etc. ECG, blood pressure, heart rate, respiratory status and lab test indexes including blood, urine, liver and kidney function, etc are all normal within 4 weeks before screening;
* No close contacts of tuberculosis;
* Subjects have not participated in other clinical drug trials or inoculated against other prophylactic and immune globulin in the nearly 3 months;
* Temperature is normal;
* Stop smoking, drinking and drinking contains caffeinated.

Exclusion Criteria:

* Health people have close contacts of TB (Tuberculosis)patients, especially excreter in 3 weeks before selection;
* Suffering from any other serious disease, e.g. during cancer treatment, autoimmune disease, progressive atherosclerosis, diabetes accompanied with complications, chronic obstructive pulmonary disease (COPD) needing oxygen therapy, acute or progressive liver or kidney disease, congestive heart failure, etc.;
* People have history of allergy, convulsions, epilepsy, cerebropathy, neurological symptoms and signs;
* Patients who have impaired or abnormal immune function, e.g. patients treated with immunosuppressor or immunopotentiator, received immunoglobulin preparation or blood products or plasma extraction outside the gastrointestinal tract in 3 months, human immunodeficiency virus or related diseases;
* Acute febrile illness and infection;
* Taking part in other clinic trials;
* Subjects have participated in any other clinical drug trials in 3 months before our clinical tests;
* Allergic constitution, e.g. patients have allergic history to two or more kinds of drugs or food, or drug components;
* Substance abuse and alcoholics ;
* Pregnant or breast feeding women;
* Mental or physical disability;
* Informed leavers;
* Any other cases that may influence the test evaluation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, Bachelor, Principal Investigator — Shanghai Public Health Clinical Center

REFERENCES:
- [Background] van Pinxteren LA, Ravn P, Agger EM, Pollock J, Andersen P. Diagnosis of tuberculosis based on the two specific antigens ESAT-6 and CFP10. Clin Diagn Lab Immunol. 2000 Mar;7(2):155-60. doi: 10.1128/CDLI.7.2.155-160.2000. PMID 10702486
- [Background] Ravn P, Munk ME, Andersen AB, Lundgren B, Lundgren JD, Nielsen LN, Kok-Jensen A, Andersen P, Weldingh K. Prospective evaluation of a whole-blood test using Mycobacterium tuberculosis-specific antigens ESAT-6 and CFP-10 for diagnosis of active tuberculosis. Clin Diagn Lab Immunol. 2005 Apr;12(4):491-6. doi: 10.1128/CDLI.12.4.491-496.2005. PMID 15817755
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738
- [Derived] Li F, Xu M, Zhou L, Xiong Y, Xia L, Fan X, Gu J, Pu J, Lu S, Wang G. Safety of Recombinant Fusion Protein ESAT6-CFP10 as a Skin Test Reagent for Tuberculosis Diagnosis: an Open-Label, Randomized, Single-Center Phase I Clinical Trial. Clin Vaccine Immunol. 2016 Sep 6;23(9):767-73. doi: 10.1128/CVI.00154-16. Print 2016 Sep. PMID 27413070
- See also: Center for drug evaluation, CFDA ,China — https://wbca.cde.org.cn/wbca/clinmain.do?method=edit&ckmIdCode=8BE5738082A97A9E5471F80B4F814FCF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In September 4, 2013, the recruitment carried out in Shanghai Public Health Clinical Center.
Groups:
- 1μg/ml ESAT6-CFP10: We get 32 healthy subjects who all meet the standard of our protocol by comprehensive check-up and asked basic medical history .32 healthy subjects are allocated four different groups according to dosages of ESAT6-CFP10 :1μg/ml ESAT6-CFP10、5μg/ml ESAT6-CFP10、10μg/ml ESAT6-CFP10、20μg/ml ESAT6-CFP10.Each dose group have six healthy subjects who are injected drug , at the same time set up two people for substitute (one male and one female) .
  Each participant intradermally inject only one dose of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 in one third site of left or right forearm palmaris .Within the same dose group two volunteer must be interval 40 minutes .
  Make sure 1μg/ml ESAT6-CFP10 group finally finished injection and observed seven days with no serious adverse reaction, then carry out 5μg/ml ESAT6-CFP10 groups .
- 5μg/ml ESAT6-CFP10: We get 32 healthy subjects who all meet the standard of our protocol by comprehensive check-up and asked basic medical history .32 healthy subjects are allocated four different groups according to dosages of ESAT6-CFP10 :1μg/ml ESAT6-CFP10、5μg/ml ESAT6-CFP10、10μg/ml ESAT6-CFP10、20μg/ml ESAT6-CFP10.Each dose group have six healthy subjects who are injected drug , at the same time set up two people for substitute (one male and one female) .
  Each participant intradermally inject only one dose of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 in one third site of left or right forearm palmaris .Within the same dose group two volunteer must be interval 40 minutes .
  Make sure 5μg/ml ESAT6-CFP10 group finally finished injection and observed seven days with no serious adverse reaction, then carry out 10μg/ml ESAT6-CFP10 groups .
- 10μg/ml ESAT6-CFP10: We get 32 healthy subjects who all meet the standard of our protocol by comprehensive check-up and asked basic medical history .32 healthy subjects are allocated four different groups according to dosages of ESAT6-CFP10 :1μg/ml ESAT6-CFP10、5μg/ml ESAT6-CFP10、10μg/ml ESAT6-CFP10、20μg/ml ESAT6-CFP10.Each dose group have six healthy subjects who are injected drug , at the same time set up two people for substitute (one male and one female) .
  Each participant intradermally inject only one dose of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 in one third site of left or right forearm palmaris .Within the same dose group two volunteer must be interval 40 minutes .
  Make sure 10μg/ml ESAT6-CFP10 group finally finished injection and observed seven days with no serious adverse reaction, then carry out 20μg/ml ESAT6-CFP10 groups .
- 20μg/ml ESAT6-CFP10: We get 32 healthy subjects who all meet the standard of our protocol by comprehensive check-up and asked basic medical history .32 healthy subjects are allocated four different groups according to dosages of ESAT6-CFP10 :1μg/ml ESAT6-CFP10、5μg/ml ESAT6-CFP10、10μg/ml ESAT6-CFP10、20μg/ml ESAT6-CFP10.Each dose group have six healthy subjects who are injected drug , at the same time set up two people for substitute (one male and one female) .
  Each participant intradermally inject only one dose of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 in one third site of left or right forearm palmaris .Within the same dose group two volunteer must be interval 40 minutes .
Period: Overall Study
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Aged from 18 to 40 years old, the male to female ratio of cases is 1:1 in each group . Body mass index should be in the range of 20 to 27 .
Groups:
- 1μg/ml ESAT6-CFP10; 5μg/ml ESAT6-CFP10; 10μg/ml ESAT6-CFP10; 20μg/ml ESAT6-CFP10: 24 healthy subjects who meet the standard of protocol are allocated four different groups according to dosages of ESAT6-CFP10 :1μg/ml Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10、5μg/ml Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10、10μg/ml Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10、20μg/ml Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10.Each dose group have six healthy subjects , at the same time set up two people for substitute (one male and one female) .
- Total: Total of all reporting groups
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.00 (3.93) | 25.63 (4.13) | 30.07 (4.00) | 27.68 (3.79) | 27.10 (3.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 12
  Male | 3 | 3 | 3 | 3 | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.32 (2.03) | 23.07 (2.05) | 22.05 (1.13) | 22.88 (2.11) | 22.58 (1.83)
height [Mean (Standard Deviation); unit: cm] | 169.17 (11.97) | 169.00 (9.67) | 163.00 (5.06) | 164.83 (11.11) | 166.50 (9.45)

OUTCOME MEASURES:

1. Primary Outcome: the Cases of Adverse Events With Participant Injection of ESAT6-CFP10
Description: The main examination items :vital signs (breathing, heart rate, blood pressure, body temperature ) of each volunteer at 15min, 30min, 1h, 2h, 4h, 8h, 24h, 48h, 72h, 96h after injection, skin reactivity (redness and/or induration) of injection sites,local reaction ( rash, pain, itching, and skin mucous membranes ) ,a variety of adverse events,routine blood,routine urine, liver and kidney function, ECG and chest X-ray films before and 7 days after intradermal injection .
Time Frame: within 7 days after the injections
Population: ESAT6-CFP10 allergen similar to TB-PPD(Tuberculin purified protein derivative ), main ingredients are protein and can cause specific skin allergy in the injection site ( such as redness, swelling, induration, blisters), besides other local reactions, is still listed as adverse events .
Measure: Number; unit: cases
Groups:
- 1μg/ml ESAT6-CFP10: Concentration of 1 ug/ml;dosage form:Injection; 0.3 ml/bottle; Intradermal injection; 0.1 ml per participants; a single dose
- 5μg/ml ESAT6-CFP10: Concentration of 5 ug/ml;dosage form:Injection; 0.3 ml/bottle; Intradermal injection; 0.1 ml per participants; a single dose
- 10μg/ml ESAT6-CFP10: Concentration of 10ug/ml;dosage form:Injection; 0.3 ml/bottle; Intradermal injection; 0.1 ml per participants; a single dose
- 20μg/ml ESAT6-CFP10: Concentration of 20 ug/ml;dosage form:Injection; 0.3 ml/bottle; Intradermal injection; 0.1 ml per participants; A single dose
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 6 | 6 | 6 | 6
cases | 3 | 1 | 0 | 0

2. Secondary Outcome: the Number of Participants Who Appear the Induration and/or Redness 2h After Application of ESAT6-CFP10
Description: We check the immune response( induration and/or redness) at 2h after application of ESAT6-CFP10 with vernier caliper. Using the standardized vernier caliper, measured transverse diameter and the longitudinal diameter of induration and/or redness in skin test parts if any participants appear induration and/or redness after application of ESAT6-CFP10.
Time Frame: within 2h after application of ESAT6-CFP10
Population: Induration and/or redness is our main immune response of ESAT6-CFP10.
Measure: Number; unit: participants
Groups:
- 10μg/ml ESAT6-CFP10: Concentration of 10 ug/ml;dosage form:Injection; 0.3 ml/bottle; Intradermal injection; 0.1 ml per participants; a single dose
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: the Number of Participants Who Appear the Induration and/or Redness 24h After Application of ESAT6-CFP10
Description: We check the immune response( induration and/or redness) at 24h after application of ESAT6-CFP10 with vernier caliper. Using the standardized vernier caliper, measured transverse diameter and the longitudinal diameter of induration and/or redness in skin test parts if any participants appear induration and/or redness after application of ESAT6-CFP10.
Time Frame: 24h after application of ESAT6-CFP10
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

4. Secondary Outcome: the Number of Participants Who Appear the Induration and/or Redness 48h After Application of ESAT6-CFP10
Description: We check the immune response( induration and/or redness) at 48h after application of ESAT6-CFP10 with vernier caliper. Using the standardized vernier caliper, measured transverse diameter and the longitudinal diameter of induration and/or redness in skin test parts if any participants appear induration and/or redness after application of ESAT6-CFP10.
Time Frame: 48h after application of ESAT6-CFP10
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

5. Secondary Outcome: the Number of Participants Who Appear the Induration and/or Redness 72h After Application of ESAT6-CFP10
Description: We check the immune response( induration and/or redness) at 72h after application of ESAT6-CFP10 with vernier caliper. Using the standardized vernier caliper, measured transverse diameter and the longitudinal diameter of induration and/or redness in skin test parts if any participants appear induration and/or redness after application of ESAT6-CFP10.
Time Frame: 72h after application of ESAT6-CFP10
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

6. Secondary Outcome: the Number of Participants Who Appear the Induration and/or Redness 96h After Application of ESAT6-CFP10
Description: We check the immune response( induration and/or redness) at 96h after application of ESAT6-CFP10 with vernier caliper. Using the standardized vernier caliper, measured transverse diameter and the longitudinal diameter of induration and/or redness in skin test parts if any participants appear induration and/or redness after application of ESAT6-CFP10.
Time Frame: 96h after application of ESAT6-CFP10
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: We collected and recorded all kinds of adverse event data within seven days after injection with ESAT6-CFP10.
Groups:
- 1μg/ml ESAT6-CFP10: Medicine Number 6 participant 24 h after test skin test, is observed local skin reactions and found subcutaneous hemorrhage ( 2 x 2 mm),48 h the subcutaneous hemorrhage is remain and becomes shallow ,72 h the subcutaneous hemorrhage is the same size and becomes lower shallow ,96 h the skin reaction has faded .This mild local skin reactions may be relevant with acupuncture of skin test , had nothing to do with experimental drugs by the judgement of principal investigator .
  Medicine Number 12 participant occurred two cases of adverse events the seventh days after skin test :respectively pregnancy and a small amount of pleural effusion on both sides .This volunteer test results of a pregnancy test paper were negative in screening period,pregnancy test result were positive the seventh days after the skin test.
- 5μg/ml ESAT6-CFP10: Medicine Number 2 participant 15 min and 30 min after skin test is observed local skin reactions and all found that scattered red dot (32 x 25 mm )appeared .After 30min each time point local skin reactions were negative .
  This mild local skin reactions may be relevant with alcohol allergy , had nothing to do with experimental drugs by the judgement of principal investigator .
- 10μg/ml ESAT6-CFP10; 20μg/ml ESAT6-CFP10: There is no adverse event.
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1μg/ml ESAT6-CFP10 (N=6) | 5μg/ml ESAT6-CFP10 (N=6) | 10μg/ml ESAT6-CFP10 (N=6) | 20μg/ml ESAT6-CFP10 (N=6)
Subcutaneous Hemorrhage Caused by Injection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
alcohol allergy caused by disinfection of the injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This volunteer test results of a pregnancy test paper were negative in screening period,pregnancy test result were positive the seventh days after the skin test.
a small amount of effusion in bilateral chest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The participant had trace pleural effusion before injection.7 days after injection found a small amount of effusion was in bilateral chest .Participant refused follow-up and not have any discomfort ,so effusion had nothing to do with drugs .

LIMITATIONS AND CAVEATS:
If the operator don't have standard measurement of transverse diameter and the vertical diameter of induration or redness ,we get unreliable data .The participant lost any follow-up will lead to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other